CLINICAL TRIAL: NCT02347488
Title: Testing a Novel Combined Endotracheal Tube Holder and Bite Guard in Neurosurgical Patients, Thoracic Surgery Patients, and Orthopedic and Neurosurgical Spine Surgery Patients.
Brief Title: Endotracheal Tube Holder and Bite Guard Research
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Nir Hoftman, M.D., MD, Associate Clinical Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-001836
Record Dates: First submitted 2015-01-08; First posted 2015-01-27 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Surgery; Anesthesia
Keywords: ETT Holder, bite guard, airway, endotracheal tube
MeSH Terms: interventions — Mouth Protectors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ETT holder and bite guard (Experimental): Participants will have endotracheal tubes secured with tape prior to having surgery, which is the current standard of care. Following the traction test and measurement of displacement, participants will have endotracheal tubes secured with a combined Haider ETT Tube Holder and Bite Guard.
  Interventions: Device: Haider ETT Tube Holder and Bite Guard; Procedure: Tape

INTERVENTIONS:
Device: Haider ETT Tube Holder and Bite Guard — Surgery patients will have endotracheal tubes secured with a novel combined endotracheal tube holder and bite guard change in ETT tip position caused by traction up to 15N was measured prior to surgery.
  Other Names: ETT Tube Holder and Bite Block
Procedure: Tape — Surgery patients will have endotracheal tubes secured with adhesive tape, as the current clinical procedure; change in ETT tip position caused by traction up to 15N measured prior to re-securing the ETT with the Haider device.

SUMMARY:
This study aims to test the effectiveness of a novel combined endotracheal tube holder and bite guard when compared with the current standard of care, tape and an oral airway.

DETAILED DESCRIPTION:
Endotracheal tubes (ETT) are secured during surgery and ICU care so that they are not accidentally removed from the airway. The position of the tip of the ETT is important and must not vary much within the trachea. The standard technique for securing an ETT is to use tape to attach it to the upper lip and face. The technique is cheap and simple, but suffers from certain drawbacks. First, the upper lip is mobile and thus even when well secured, the tube can move within the trachea due to this mobility. Second, conditions on the face such as sweating, drooling, facial hair, skin flaking or breakdown, all interfere with the ability of the tape to adhere, thus reducing its efficacy. Furthermore, the tape itself can irritate and or injure the facial skin. The adhesive irritates skin and certain patients are allergic to these substances. Also, removing the tape can physically damage the skin, especially if the skin is vulnerable to sheer forces (such as elderly patients or patients on systemic steroids).

Patients that are intubated often need a bite block or bite guard inserted into their mouths. This serves two main purposes: 1) to prevent the patient from biting the ETT and occluding airflow, 2) to prevent the patient from biting their tongue, cheek, or lips causing injury. Furthermore, endoscopic procedures are often performed on intubated patients and thus a bite block is needed to protect the delicate instrument from being bitten and damaged. For these reasons, many providers will insert bite blocks into the mouths of intubated patients. Many such devices exist on the market, but the most commonly used is the Guedel oral airway. This device is actually designed to increase airway patency during mask ventilation, and long term use of this device as a bite block has been linked to numerous complications including: 1)tongue swelling, often compromising the airway patency, 2) tooth damage, and 3)lip injury. Because of these shortcomings, specific ETT bite blocks have been developed, and some of these even double as an ETT securing device. However, these are usually made of hard, stiff materials that in and of themselves can injure the delicate oral structures. In summation, no single device that both serves as an ergonomic ETT holder and bite block has been successfully developed and marketed, and therefore the standard of care remains tape plus an oral airway.

The Haider airway is a combination ETT holder-securing device and bite block. Made of soft silicone rubber, the device was engineered from the ground up to serve those purposes with safety and comfort in mind. The device is FDA approved and in a pre-marketing trials phase to determine the efficacy of the product in specific clinical scenarios. Our institution has been tasked with testing the device in clinical scenarios where tape + oral airway has been historically problematic. We plan to compare this new device to tape + oral airway, the current standard of care in neurosurgical patients in the supine position. We hypothesize the device will be superior to the standard of care in both efficacy and patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* General anesthesia requiring oral endotracheal intubation in the prone position for the duration of surgery (head secured in a foam head holder, horseshoe frame, or Mayfield pins).
* General anesthesia for neurosurgery requiring oral endotracheal intubation, supine or slight lateral bump position for the duration of surgery. (Special emphasis will be placed on including patients who will undergo motor evoked potentials, and thus will not be paralyzed during the surgery).
* General anesthesia requiring oral endotracheal intubation with a left sided double-lumen endotracheal tube for lung isolation, lateral position for the duration of surgery.

Exclusion Criteria:

* Dentition issues (loose teeth, missing teeth)
* Temporomandibular joint disease
* Maxillofacial abnormalities (deformities of the jaw, lips, tongue)
* Surgical procedures involving the teeth, lips, jaw
* History of asthma or bronchospasm
* Immunosuppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nir Hoftman, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Tape, Followed by ETT Holder and Bite Guard: Tape: Surgery patients had endotracheal tubes secured with adhesive tape, as the current clinical procedure; change in ETT tip position caused by traction up to 15N measured prior to re-securing the ETT with the Haider device.
  Haider ETT Tube Holder and Bite Guard: Surgery patients then had endotracheal tubes secured with a novel combined endotracheal tube holder and bite guard; change in ETT tip position caused by traction up to 15N measured prior to surgery.
Period: Overall Study
Arm/Group | Tape, Followed by ETT Holder and Bite Guard
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tape, Followed by ETT Holder and Bite Guard
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 55.4 [22 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in ETT Position
Description: The ability of the securing device to resist endotracheal tube dislodgement under axial strain for patients in the supine position was measured. The endotracheal tube, once secured with either tape or the Haider airway device, encountered an axial force to simulate the endotracheal tube being pulled from the mouth. The force increased over approximately 5 seconds until the target of 15 N was reached or until the principal investigator deemed that the force be aborted to prevent possible tracheal extubation. The change in position, measured in cm, was recorded.
Time Frame: 5 minutes after intubation (which occurs at the beginning of the anesthesia about 2-5 minutes after the patient goes to sleep).
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Adhesive Tape: Participants had endotracheal tubes secured with tape prior to having surgery, which is the current standard of care. Following the traction test and measurement of ETT tip position displacement, endotracheal tubes were re-secured with a combined Haider ETT Tube Holder and Bite Guard.
- Haider ETT Tube Holder: Following the traction test and measurement of taped ETT tip position displacement, endotracheal tubes were re-secured with a combined Haider ETT Tube Holder and Bite Guard.
Arm/Group | Adhesive Tape | Haider ETT Tube Holder
Number analyzed (Participants) | 30 | 30
centimeters | 3.4 (1.8) | 0.3 (0.6)
Statistical Analysis 1: Comparison: Adhesive Tape vs Haider ETT Tube Holder; Average displacement difference in cm, tape vs. tube-holder. 17 participants was the estimated enrollment needed to detect a difference of 1 SD from the mean between the 2 fixation techniques at 80% power; additional enrollment was included to increase the power of results and to include a larger variety of patients undergoing different surgical procedures; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [2.88 to 3.32], Standard Deviation 1.8

2. Secondary Outcome: Participants With Irritation or Minor Injury to the Face and Oral Structures Likely Attributable to the Study Device
Description: The patients were examined after surgery (both immediately after surgery and at the end of the recovery room period) to determine if the patient suffered any irritation or minor injury to the face and oral structures. The patients were asked to fill out a questionnaire after recovery with questions about their overall experience with specific relation to any irritation and/or minor trauma to their face, oral structures, throat, jaw, and temporomandibular joint.
Time Frame: Immediately after surgery and 1-3 days following surgery, before discharge.
Population: 29 patients returned the survey (one patient was aphasic post-op and could not compete the survey)
Measure: Count of Participants; unit: Participants
Arm/Group | Tape, Followed by ETT Holder and Bite Guard
Number analyzed (Participants) | 29
Participants | 2

3. Secondary Outcome: Clinically Significant Movement
Description: Number of participants experiencing ETT movement >1cm under each fixation technique
Time Frame: 5 minutes after intubation (which occurs at the very beginning of the anesthesia about 2-5 minutes after the patient goes to sleep)
Measure: Count of Participants; unit: Participants
Arm/Group | Adhesive Tape | Haider ETT Tube Holder
Number analyzed (Participants) | 30 | 30
Participants | 29 | 1

4. Secondary Outcome: Potentially High Extubation Risk
Description: Number of participants experiencing ETT movement >4cm under each fixation technique
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Adhesive Tape | Haider ETT Tube Holder
Number analyzed (Participants) | 30 | 30
Participants | 9 | 0

ADVERSE EVENTS:
Time Frame: Immediately after surgery and up to 1-3 days following surgery, before discharge.
Description: Unfavorable findings were recorded as adverse events in this study only if severe, unexpected, or considered to have been attributable to use of the study device.
Groups:
- Tape, Followed by ETT Holder and Bite Guard: Tape: Surgery patients had endotracheal tubes secured with adhesive tape, as the current clinical procedure; change in ETT tip position caused by traction up to 15N measured prior to re-securing the ETT with the Haider device.
  Haider ETT Tube Holder and Bite Guard: Surgery patients then had endotracheal tubes secured with a novel combined endotracheal tube holder and bite guard; change in ETT tip position caused by traction up to 15N measured prior to surgery.
  Adverse events were not reported "per arm" because surgery patients were assessed for adverse events after experiencing both methods.
Arm/Group | Tape, Followed by ETT Holder and Bite Guard
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tape, Followed by ETT Holder and Bite Guard (N=30)
Mild discomfort of the gum (Gastrointestinal disorders) | 1 (1)
minor abrasion of the tongue frenulum (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes